CLINICAL TRIAL: NCT04620122
Title: Adiyaman University
Brief Title: Effects of Progressive Muscle Relaxation Training With Music Therapy on Sleep Quality and Trait Anger/Anger Expression Style of Patients at Community Mental Health Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Ceyda Başoğul, Principal Investigator, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/4-1
Record Dates: First submitted 2020-11-03; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Sleep; Anger; Psychiatric Disorder
Keywords: sleep quality; Anger; Psychiatric Disorder; therapy
MeSH Terms: conditions — Mental Disorders; Sleep Initiation and Maintenance Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Progressive Muscle Relaxation Training and Music Therapy are applied to the intervention group.
  Interventions: Other: Progressive Muscle Relaxation Training and Music Therapy
- control group (No Intervention): No intervention is applied to the control group.

INTERVENTIONS:
Other: Progressive Muscle Relaxation Training and Music Therapy — Progressive Muscle Relaxation Training and Music Therapy have applied to the participants two sessions for a week during two months.
  Arms: intervention group

SUMMARY:
Aim: The aim of the study was to examine the effects of progressive muscle relaxation training with music therapy on sleep quality, trait anger, and anger expression style of patients at the community mental health center.

Method: The study is conducted as the pretest-posttest control group design. The study population consisted of chronic psychiatric patients who continue in a Community Mental Health Center located in southeastern Turkey. The days when the participants came to the Community Mental Health Center were selected and the participants divided into two groups as an intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* Having a chronic psychiatric diagnosis according to DSM-V diagnostic criteria,
* Open and cooperate for communication,
* living in the city center,
* age was between 18-60

Exclusion Criteria:

* Patients who have just started the Community Mental Health Center
* patients diagnosed with axis 1,
* patients diagnosed with mental retardation,
* patients with drug or alcohol addiction,
* patients diagnosed with organic brain syndrome,

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 2 minutes
  PSQI is a self-report scale that evaluates sleep quality and disturbance over a one-month period. PSQI was developed by Buysse et al. (1989). The validity and reliability study of PSQI in our country was conducted by Ağargün et al. (1996) (Cronbach's alpha = 0.80).
The Trait Anger/Anger Expression Inventory | 2 minutes
  It was developed by Spielberger et al. (1983). Turkish adaptation of the scale was made by Özer and Kadir (1994). The first 10 items of the scale measure trait anger and the next 24 items measure anger expression styles.

CONTACTS AND LOCATIONS:
Locations (1):
- Community Mental Health Center, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Icel S, Basogul C. Effects of progressive muscle relaxation training with music therapy on sleep and anger of patients at Community Mental Health Center. Complement Ther Clin Pract. 2021 May;43:101338. doi: 10.1016/j.ctcp.2021.101338. Epub 2021 Feb 19. PMID 33639518